CLINICAL TRIAL: NCT02598206
Title: A Phase 1, Randomized, Open Label, Single Dose, 2-period Crossover Study To Evaluate Food Effect On The Pharmacokinetics Of Pf-04136309 In Healthy Subjects
Brief Title: Food Effect Study PF-04136309
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A9421019; 2015-003649-24 (EudraCT Number)
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Healthy
Keywords: food effect; healthy volunteers; pharmacokinetics; CCR2i
MeSH Terms: interventions — PF-04136309

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental 1 (Experimental): All subjects will receive 2 treatments in one of the indicated sequence orders:
  A - B B - A
  Interventions: Drug: PF-04136309

INTERVENTIONS:
Drug: PF-04136309 — Treatment A (n=18): a single dose of 1000 mg PF 04136309 will be administered in a fasted state as 8 × 125 mg Tablets.
  Treatment B (n=18): a single dose of 1000 mg PF-04136309 will be administered with a high fat breakfast as 8 × 125 mg Tablets.

SUMMARY:
The purpose of this study is to evaluate the effect of food intake on PF-04136309 pharmacokinetics (PK) following a single dose at 1000 mg.

DETAILED DESCRIPTION:
The present study will be conducted in healthy adult subjects. The single dose of 1000 mg has been shown to be safe in a previous study in healthy subjects. To evaluate the effect of food on PF-04136309 PK at the dose of 1000 mg, which is the maximum dose that may be evaluated in the multiple dose setting in patients, will provide information to guide the dose administration in regards to food intake at relevant therapeutic dose levels for further studies in patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of non childbearing potential, who at the time of screening are between the ages of 45 55, and/or male subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Subjects who are smoking, or with evidence of disease, conditions affecting absorption, treatment with other investigational drug within 30 days, history of regular alcohol consumption, use of prescription, nonprescription drugs and dietary supplement within 7 days, or blood donation of 500 mL within 56 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve from time Zero to Extrapolated Infinite Time (AUC[0-inf]). | 0(pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours (hrs) post-PF-04136309 dose
  AUC(0-inf)=Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (o-inf). It is obtained from AUC (0-t) plus AUC (t-inf).
Maximum Plasma Concentration [Cmax] | 0(pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hrs post PF-04136309 dose

SECONDARY OUTCOMES:
Area Under the Curve from Time Zero to Last Quantifiable Concentration (AUClast) | 0(pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hrs post PF-04136309
  Area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration (AUClast).
Time to Reach maximum Observed Plasma Concentration (Tmax) | 0(pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hrs post PF-04136309 dose
  Time for Cmax
Plasma Decay Half Life (t1/2) | 0(pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hrs post PF-04136309
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Apparent Oral Clearance (CL/F) | 0(pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hrs post-PF-04136309 dose
  Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Apparent Volume of Distribution (Vz/F) | 0(pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hrs post PF-04136309 dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9421019&StudyName=A%20Phase%20I%20Randomized%20Open%20Label%2C%20Single%20Dose%2C%202-period%20Crossover%20Study%20To%20Evaluate%20Food%20Effect%20On%20The%20Pharmacokinetics%20Of%20Pf-04136309%20In%20Healthy%20Volunteers.